CLINICAL TRIAL: NCT06325332
Title: BEYFORTUS™ (Nirsevimab) Effectiveness Against Medically-Attended RSV Events in Infants (BEAR Study)
Acronym: BEAR
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: RSV00080
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Virus
Keywords: RSV
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Cohort 1: Nirsevimab-Exposed Cohort: Full-term (born ≥ 37 weeks gestational age) infants born on or after 01 April 2023, without a high-risk condition, who receive nirsevimab before or during their first RSV season per recommendations, ie, before or during the 2023-2024 RSV season.
  Interventions: Other: Nirsevimab
- Cohort 2: Comparator Cohort: Full-term (born ≥ 37 weeks gestational age) infants born on or after 01 April 2023, without a high-risk condition, who do not receive nirsevimab before or during the 2023-2024 RSV season.
- Cohort 3: Historical Control Cohort: Full-term (born ≥ 37 weeks gestational age) infants without a high-risk condition from previous RSV seasons 2016-2017, 2017-2018, 2018-2019, 2019-2020, and 2022-2023. The 2020-2021 and 2021-2022 seasons are excluded due to low circulation of RSV during the COVID-19 pandemic. Historical seasons' data are intended for descriptive purpose only, to contextualize the impact of the treatment during the 2023-2024 season.
- Cohort 4: Infant Cohort with High-Risk Conditions: Infants born < 37 weeks gestational age and those diagnosed with a high-risk condition between birth and the end of the observation period (regardless of gestational age at birth), will be considered infants with high-risk conditions. Infants with high-risk conditions will be excluded from Cohort 1, Cohort 2, and Cohort 3. Descriptive statistics will be separately assessed for this high-risk cohort.

INTERVENTIONS:
Other: Nirsevimab — Route of Administration: Intramuscular Pharmaceutical Form: Solution for injection
  Other Names: Beyfortus™
  Groups: Cohort 1: Nirsevimab-Exposed Cohort

SUMMARY:
The primary objectives of the study are: To estimate the effectiveness of nirsevimab against polymerase chain reaction (PCR)-confirmed RSV (1) lower respiratory tract (LRTD) and (2) related medical encounters.

the secondary objectives are:

1. To estimate the effectiveness of nirsevimab against medical encounters with a respiratory related diagnosis.
2. To estimate the effectiveness of nirsevimab against medical encounters with an LRTD diagnosis.
3. To estimate the impact of nirsevimab on PCR-confirmed RSV.
4. To estimate the impact of nirsevimab on medical encounters with an otitis media diagnosis.
5. To estimate the impact of nirsevimab on antibiotic prescription.

ELIGIBILITY:
Inclusion Criteria:

* The Kaiser Permanente Northern California, USA (KPNC) member born on or after 01 April 2023 for Cohort 1 and Cohort 2.
* Eligible to receive nirsevimab as defined by the product indication.
* KPNC infants entering their first RSV season.

Exclusion Criteria:

* Mother was administered an RSV vaccine during her pregnancy with the infant participant.
* Mother of infant participant was not a KPNC member during pregnancy.
* Mother did not deliver the infant participant at a KPNC facility.
* Infant receipt of other RSV pre-exposure prophylaxis (ie, Palivizumab).

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study is an observational, retrospective cohort study designed to evaluate the effectiveness of nirsevimab to prevent RSV-confirmed respiratory-related medical encounters and health care utilization in infants entering their first RSV season compared to no treatment in the United States.
  The source population is infants ≥ 37 weeks gestational age and aged 0 to 12 months (calendar age) entering their first RSV season and without significant medical history. There is also a high-risk infant population with infants < 37 WGA and aged 0 to 12 months (calendar age), entering their first RSV season and infants ≥ 37 weeks with significant medical history diagnosed at birth up to the end of the observation period (ie, 30 April 2024). The study will aim to enroll approximately 33,000 infants.
Sampling Method: Probability Sample
Enrollment: 49680 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of first episodes of polymerase chain reaction (PCR)-confirmed RSV with an lower respiratory tract disease (LRTD) | Approximately 6 months
  Incidence of first episodes of polymerase chain reaction (PCR)-confirmed RSV with an lower respiratory tract disease (LRTD) diagnosis identified using International Classification of Diseases, Tenth Revision (ICD)
Number of medical encounters associated with the first episode of PCR-confirmed RSV with a LRTD diagnosis | Approximately 6 months
  Number of medical encounters associated with the first episode of PCR-confirmed RSV with a LRTD diagnosis identified using ICD-10 codes: outpatient (OP) visits, emergency department (ED) visits, inpatient (IP) hospitalizations or intensive care unit (ICU) hospitalizations.

SECONDARY OUTCOMES:
Number of respiratory-related medical encounters | Approximately 6 months
  Number of respiratory-related medical encounters (ie, Outpatient visits, Emergency department visits, In patient hospitalizations, and Intensive care unit hospitalizations) by ICD-10 codes.
Number of respiratory-related medical encounters for LRTD by ICD-10 codes | Approximately 6 months
  Number of respiratory-related medical encounters for LRTD by ICD-10 codes.
Incidence of PCR-confirmed RSV (first occurrence of season) | Approximately 6 months
  Incidence of PCR-confirmed RSV (first occurrence of season).
Number of medical encounters for otitis media by ICD-10 codes | Approximately 6 months
  Number of medical encounters for otitis media by ICD-10 codes.
Number of antibiotic prescriptions by National Drug Code (NDC) codes | Approximately 6 months
  Number of antibiotic prescriptions by NDC codes.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northern California: Site number 0001, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org